CLINICAL TRIAL: NCT03182972
Title: Intervention Study on Medication Reconciliation Among Pharmacists in Two Tertiary Hospitals in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, AKINNIYI AKINBIYI AJE, Lecturer II, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MR/UCH/FMC/73247
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Intervention Study
Keywords: intervention study; medication reconciliation; pharmacists; Nigeria; Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Medication Reconciliation

STUDY DESIGN:
Intervention Model Description: University College Hospital, Ibadan will serve as the intervention group while University of Ilorin Teaching Hospital, Ilorin will serve as the control group.
Who Masked: Participant, Care Provider
Masking Description: Both the patients and the pharmacists recruited for the study will not be informed whether they are in the control or intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Seminar presentation will be done using the followings:
  1. Power point presentation on the following topics as it relates to medication reconciliation:
     1. Communication skill (with patients and also with other members of the healthcare team)
     2. Documentation of pharmaceutical care activities
     3. Medication history taking
     4. Drug therapy problems
     5. Medication reconciliation practice
  2. Case studies on medication reconciliation
  3. Role plays on medication reconciliation
  Interventions: Other: Medication reconciliation
- Control arm (No Intervention): Control group

INTERVENTIONS:
Other: Medication reconciliation — Pre-post intervention
  Arms: Intervention arm

SUMMARY:
This study will assess the current practice of medication reconciliation among pharmacists in the selected institutions with a view to making an intervention to address gaps discovered

DETAILED DESCRIPTION:
Background information garnering will be done among the pharmacists in the two selected hospitals to collect data on current practice of medication reconciliation. Focus group discussion will be done in the intervention group so as to identify peculiarities of their practice and to provide the best approach to carrying out the intervention. Diabetes and hypertensive patients in medical outpatient clinic will be interviewed in order to assess current practice of medication reconciliation.

Intervention will be channeled towards addressing gaps discovered. University College Hospital, Ibadan, Oyo State will be the intervention group, while University of Ilorin Teaching Hospital, Kwara State will be the control group.

The effect of the intervention will be measured over time to ensure that medication reconciliation is implemented in the selected institutions.

ELIGIBILITY:
Inclusion Criteria:

* Participant has diabetes and/or hypertension
* Registered pharmacists in the selected institutions

Exclusion Criteria:

* Participants that are neither diabetic nor hypertensive
* Unregistered pharmacists in the selected institutions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Medication reconciliation: Percentage unreconciled medications | 3 months
  Percentage unreconciled medications

CONTACTS AND LOCATIONS:
Overall Officials: TITILAYO O FAKEYE, PhD, Study Director — University of Ibadan
Locations (2):
- Nigeria (2):
  - University of Ilorin Teaching Hospital, Ilorin, Kwara State
  - University College Hospital, Ibadan, Oyo State

IPD SHARING:
Plan to Share IPD: Yes